CLINICAL TRIAL: NCT01275209
Title: A Phase Ib, Multicenter, Open-label Study of HCD122 Administered Intravenously in Combination With Bendamustine in Patients With CD40+ Follicular Lymphoma Who Are Refractory to Rituximab
Brief Title: Study of HCD122 (Lucatumumab) and Bendamustine Combination Therapy in CD40+ Rituximab-refractory Follicular Lymphoma
Acronym: LIFT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHCD122A2104; 2010-022350-17 (EudraCT Number)
Record Dates: First submitted 2011-01-10; First posted 2011-01-12 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2012-12

CONDITIONS: Follicular Lymphoma
Keywords: HCD122; Lucatumumab; CD40; Follicular Lymphoma; Non-Hodgkin's Lymphoma; Antibody
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — lucatumumab

ARMS (1):
- HCD122 (Experimental)
  Interventions: Drug: HCD122

INTERVENTIONS:
Drug: HCD122
  Other Names: Lucatumumab

SUMMARY:
This study will assess the safety and efficacy of HCD122 (Lucatumumab) when combined with bendamustine in patients with follicular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of follicular lymphoma, according to the Revised European American Lymphoma/World Health Organization [REAL/WHO] classification
* Documented CD40+ follicular lymphoma
* Measurable lesion
* Refractory to rituximab
* Prior treatment with at least 1 chemotherapeutic regimen
* 18 years or older
* WHO Performance Status grade 0, 1, or 2
* Life expectancy > 3 months
* Obtained written informed consent

Exclusion Criteria:

* Grade 3b follicular lymphoma or evidence that the indolent lymphoma has transformed to aggressive lymphoma (i.e. DLBCL)
* History of another primary malignancy that is currently clinically significant or currently requires active intervention
* Prior allogeneic stem cell transplantation
* Prior anaphylactic or other severe infusion reaction such that the patient is unable to tolerate human immunoglobulin or monoclonal antibody administration
* Impaired cardiac function or clinically significant cardiac disease
* History of acute or chronic pancreatitis, surgery of the pancreas, or any risk factors that may increase the risk of pancreatitis
* History of an active infection (viral, bacterial, or fungal) requiring systemic therapy within 28 days before study treatment.
* Known diagnosis of human immunodeficiency virus (HIV) infection
* Evidence of previous hepatitis viral infection such as hepatitis B or hepatitis C
* Ongoing corticosteroid use (>10 mg/day prednisone or equivalent)
* Pregnant or nursing (lactating) women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Incidence rate of dose-limiting toxicities and adverse events | 2 years

SECONDARY OUTCOMES:
Response rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (4):
  - Dana Farber Cancer Institute SC-5, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute Dept.of KarmanosCancerInst (6), Detroit, Michigan
  - Duke University Medical Center Duke Hem & Onc, Durham, North Carolina
  - Sarah Cannon Research Institute SC - 2, Chattanooga, Tennessee
- Novartis Investigative Site, Prahran, Victoria, Australia
- Belgium (2):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Paris, France
- Novartis Investigative Site, Torino, TO, Italy
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid

REFERENCES:
- See also: Results for CHCD122A2104 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8184